CLINICAL TRIAL: NCT05186883
Title: Treatment of Postoperative Hypoparathyroidism Using Cultured Allogenic Parathyroid Cells
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_Parathyr
Record Dates: First submitted 2021-12-01; First posted 2022-01-11 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Hypoparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with allogenic parathyroid cells (Experimental): Patients with postoperative hypoparathyroidism receiving standard treatment and allogenic parathyroid cells
  Interventions: Biological: Allogenic parathyroid cells; Other: Standard treatment according to the Clinical protocols
- Control (Active Comparator): Patients with postoperative hypoparathyroidism receiving standard treatment
  Interventions: Other: Standard treatment according to the Clinical protocols

INTERVENTIONS:
Biological: Allogenic parathyroid cells — Allogenic parathyroid cells
  Arms: Treatment with allogenic parathyroid cells
Other: Standard treatment according to the Clinical protocols — Standard treatment of postoperative hypoparathyroidism according to the Clinical protocols

SUMMARY:
The idea of the project is to develop a method of treatment of postoperative hypoparathyroidism using cultured allogenic parathyroid cells.

DETAILED DESCRIPTION:
The cells will be isolated and cultured from the parathyroid gland of brain-dead organ donors. Cells will be tested for the immunophenotype, viability, sterility and the production of parathyroid hormone. Cells will be co-cultured with the patients T-cells and the expression of perforin and granzyme B proteins will be assayed as well as the apoptosis/viability of parathyroid cells. Prepared cells will be used to treat the patients with postoperative hypoparathyroidism. The safety, tolerability and clinical efficacy will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of postoperative hypoparathyroidism
* Decreased PTH concentrations in blood serum
* The patient can read, understand, follow the examination procedures and complete, if necessary, the required documentation
* Written informed consent

Exclusion Criteria:

* The presence of any malignant tumor within the last 5 years
* Acute or chronic diseases in the stage of decompensation
* Chronic infectious diseases: HIV, viral hepatitis B, C, tuberculosis
* Patients who are pregnant, breastfeeding, or fertile patients who are not using adequate contraceptive methods
* Chronic and protracted mental disorders, all diseases with the presence of the syndrome of dependence on alcohol, drugs and psychoactive substances, any other condition that makes the patient unable to understand the nature, extent and possible consequences of the study or, in the opinion of the researcher, prevents the patient from observing and performing protocol
* Patients are unable or unwilling to give written informed consent and / or follow research procedures
* Any other medical condition that, in the opinion of the investigator, may be associated with an increased risk to the patient or may affect the outcome or evaluation of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PTH in blood serum | 3 month
  The concentration of PTH in blood serum
PTH in blood serum | 6 month
  The concentration of PTH in blood serum
PTH in blood serum | 1 year
  The concentration of PTH in blood serum
Adverse effects associated with the therapy | 1 month
  Determination of adverse effects associated with the therapy
Adverse effects associated with the therapy | 1 year
  Determination of adverse effects associated with the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Hancharou, Dr, Study Director — the Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus; Stanislav Treatiak, Prof, Study Director — Belarusian State Medical University; Andrei Bolshov, Dr, Principal Investigator — Belarusian State Medical University

IPD SHARING:
Plan to Share IPD: No